# TITLE: Program for the comprehensive neurocognitive treatment of excess weight (TRAINEP)

**Code:** RTI2018-098771-B-I00

**Date:** May 21, 2021

### TITLE: Program for the comprehensive neurocognitive treatment of excess weight (TRAINEP)

Code: RTI2018-098771-B-I00

Principal researchers: Raquel Vilar-López and Alfonso Caracuel-Romero

Email: rvilar@ugr.es, acaracuel@ugr.es

Please read this information carefully: Your voluntary participation in a research project is requested. Before participating in the study, please read the information below and ask as many questions as you need to make sure you understand what your participation entails.

#### Information about the study and your participation

#### What is the objective of the study?

The objective of this study is to determine the effectiveness of a program for the treatment of excess weight. This study is directed by Raquel Vilar López and Alfonso Caracuel Romero, and their collaborating team. The study is based at the Mind, Brain and Behavior Research Center (CIMCYC), belonging to the University of Granada, and located on the Cartuja Campus (between the faculties of Psychology and Pharmacy).

#### What procedures will I carry out?

This study includes assessments and interventions sessions. All sessions will be online. In the evaluations you will perform different tasks (through the computer and/or mobile phone) to measure different aspects related to your way of eating, exercise and physical habits, and psychological aspects (such as impulsivity and personality). Participants will be assigned to different groups of interventions on eating habits and physical exercise. In total, the study consists of 12 sessions between assessments and interventions, which will be carried out at different times over 8 months. All sessions will have a group format, with a maximum of 6 participants.

#### Potential problems participating in the study

The activities of the various assessment and intervention sessions are not expected to imply any inconvenience for the participants, beyond the exhaustion they may feel from paying attention while performing the tasks.

#### Is there any benefit from participating in the study?

Participating in the study may have benefits related to improving healthy lifestyle habits (diet and exercise), and therefore you may reduce your body weight. In addition, your participation will provide scientific insights that will help improve the design of treatments for people with excess weight.

#### Confidentiality

The personal data required (age, sex, health data ...) are necessary to meet the objectives of the study. Any personal information that may be identifiable will be kept and processed by computerized means under secure conditions. To protect your privacy, the information collected about you will be tagged with an alphanumeric code. Your results will be stored in electronic format, without identifying you name, and will be used only within the context of the project. The results derived from this study can be published in a scientific

journal or congress, always maintaining the commitment of anonymity and confidentiality. Access to this data is restricted to our research team. During the study you may at any time exercise your right of access, rectification, cancellation and opposition to your data before the responsible researcher, as established by Royal Decree 1720/2007, Organic Law 3/2018 on Protection of Personal Data and guarantee of digital rights, and European directive 2002/58/CE.

#### **Study participation agreement**

This sheet contains information so that you can decide if you want to participate in this study. If you have any questions that remain unanswered, please ask the study manager before signing this form. You can contact the main researchers of the project, Raquel Vilar López and Alfonso Caracuel Romero, through email rvilar@ugr.es and acaracuel@ugr.es or by phone 958 241 982 and 958 242 948.

Participation in this study is voluntary, and you will have the possibility to revoke your consent at any time and without having to give explanations. You do not have to participate in the study if you do not want to. If you finally decide to participate, you will receive a copy to keep this information.

### **INFORMED CONSENT**

## TITLE: Program for the comprehensive neurocognitive treatment of excess weight (TRAINEP)

| Name and surname |
|---|
| ID number |
| I have spoken with the professional responsible for the study |
| I have been invited to participate voluntarily in this study by the research team of the TRAINEP project. I agree to participate in this study, and I have made this decision freely after reading the information sheet that has been provided to me. I have had the opportunity to ask all the questions about the study that I have considered appropriate, and I have received enough information about the study. I understand that I can withdraw this consent and leave the study at any time, without having to give explanations and without receiving a penalty for doing so. I freely give my consent to participate in the study. |
| Date: |
| Signature of the participant: |
| Name of the responsible researchers: Raquel Vilar López and Alfonso Caracuel Romero |
| DNI of the responsible researchers: 46898000B and 52363377J |
| Signature of the responsible investigators: |